CLINICAL TRIAL: NCT02069457
Title: Prevalence and Predictive Factors of Portal Vein Thrombosis in Patients With Cirrhosis
Status: Completed | Type: Observational
Sponsor: Jia Ji-Dong (Other)
Responsible Party: Sponsor-Investigator, Jia Ji-Dong, Director of liver research center, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Other Study IDs: BJFH20140220
Record Dates: First submitted 2014-02-20; First posted 2014-02-24 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Liver Cirrhosis; Portal Vein Thrombosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Several studies have confirmed that patients with cirrhosis possess an imbalance in procoagulant versus anticoagulant activity due to increased factor VIII and decreased protein C. Moreover, in the last two decades there has been an increased recognition that not only bleeding but also thrombosis complicates the clinical course of cirrhosis. The prevalence and pathogenesis of portal vein thrombosis (PVT) in patients with cirrhosis without hepatocellular carcinoma are not clearly defined. The Aim of this study is to assess the prevalence of portal vein thrombosis in patients with cirrhosis without hepatocellular carcinoma, and to prospectively assess the risk factors, outcome, and prognosis in these patients. The investigators plan to enroll two hundred patients with liver cirrhosis. The patients are going to follow up for one year and evaluate at baseline and every 6 months by liver function tests, coagulation test, upper abdomen ultrasound. All relevant clinical events will be evaluated at every follow up.

ELIGIBILITY:
Inclusion Criteria:

Cirrhosis of any etiology and severity, Aged 18-80 years, Signed Informed Consent.

Exclusion Criteria:

Hepatocellular carcinoma, other intrahepatic/extrahepatic cancers, documented history of congenital coagulation disorders, pregnancy, human immunodeficiency virus (HIV) positivity, recent (<7 d) transfusion with blood products, use of anticoagulant/antiaggregation drugs in the past 10 d.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhosis of any etiology and severity
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Presence of portal vein thrombosis | 6 months
  To estimate the prevalence of PVT evaluated by US in a cohort of patients with liver cirrhosis of any etiology and severity.

SECONDARY OUTCOMES:
Cirrhosis Complications | 1 year
  Occurrence of digestive or other bleeding complications; Occurence of other cirrhosis-related complications ( onset or progression of oesophageal varices, ascites or refractory ascites, hepatic encephalopathy, onset of liver cancer, infections, spontaneous bacterial peritonitis, onset of hepato-renal or hepato-pulmonary syndrome)
Incidence of portal vein thrombosis | 1 year
  To estimate the incidence of new onset PVT evaluated by US in a cohort of patients with cirrhosis.
mortality | 1 year
  Overall mortality in a cohort of patients with cirrhosis without HCC

CONTACTS AND LOCATIONS:
Overall Officials: Jidong Jia, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China